CLINICAL TRIAL: NCT03311867
Title: Prolene Versus Ethibond for Cervical Cerclage
Acronym: PECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Meike Schuster, Assistant Professor, Rutgers University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PECC
Record Dates: First submitted 2017-10-02; First posted 2017-10-17 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cervical Incompetence
MeSH Terms: conditions — Uterine Cervical Incompetence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Braided Suture (Active Comparator): Patient in this group will have a cerclage with ethibond suture material
  Interventions: Other: Ethibond Suture
- Non- Braided Suture (Active Comparator): Patient in this group will have a cerclage with prolene suture material
  Interventions: Other: Prolene Suture

INTERVENTIONS:
Other: Ethibond Suture — Cerclage placement with ethibond
  Arms: Braided Suture
Other: Prolene Suture — Cerclage placement with prolene
  Arms: Non- Braided Suture

SUMMARY:
The purpose of the proposed study is to examine the relationship between cerclage suture material of Ethibond and Prolene and its effect on the vaginal microbiome in a prospective randomized control trial. Ethibond is another commonly used suture material for performing cervical cerclage that shares some characteristics with previously studied suture materials. It is braided like the Mersilene, but thinner like the monofilament Prolene. The investigators will study whether Ethibond causes the vaginal microbiome to be adversely affected like Mersilene or whether there is a healthy microbiome like Prolene. This study will allow the investigators to determine whether it is advisable to continue to use Ethibond for cervical cerclage in clinical practice, or whether obstetricians should avoid its use as now done with Mersilene.

ELIGIBILITY:
Inclusion Criteria:

* Greater than18 years of age
* Singleton pregnancy
* History of preterm delivery between 17 0/7 weeks - 33 4/7 weeks with painless cervical

dilation or cervical insufficiency

Exclusion Criteria:

* younger than 18 years of age
* multiple gestation
* iatrogenic preterm delivery
* pregnancies with fetal anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal Microbiome | At time of cerclage placement (11-14 wks gestation) and cerclage removal (35-36 weeks gestation)
  16S rRNA gene sequencing will be performed
Change in Vaginal Cytokine Expression | At time of cerclage placement (11-14 wks gestation) and cerclage removal (35-36 weeks gestation)
  Cytokine analysis will be performed

SECONDARY OUTCOMES:
Rate of preterm birth | Delivery between 24-26 weeks gestation
  The investigators will follow patients through their pregnancy and observe if suture material is related to increased preterm birth

CONTACTS AND LOCATIONS:
Overall Officials: Meike Schuster, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - Division of Maternal Fetal Medicine, New Brunswick, New Jersey
  - High Risk Obstetrics Clinic, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jayakumaran J, Angras K, Wang B, Paglia MJ, Rosen T, Schuster M. Monofilament vs multifilament suture for cervical cerclage: a multicenter randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Feb;5(2):100823. doi: 10.1016/j.ajogmf.2022.100823. Epub 2022 Dec 2. No abstract available. PMID 36464242